CLINICAL TRIAL: NCT00266045
Title: A Multicentre, Prospective, Observational Study on the Predictive Role for Recurrence of D-dimer Levels Measured During and After Anticoagulation in Patients With a First Venous Thromboembolism Episode (the PROLONG-II Study)
Brief Title: D-dimer Levels During and After Anticoagulation in Patients With a Previous Venous Thromboembolism: Effects on the Risk of Recurrence
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Italian Federation of Anticoagulation Clinics (FCSA) (Unknown)
Responsible Party: Principal Investigator, GUALTIERO PALARETI, Prof. Gualtiero Palareti, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: PROLONG-TWO STUDY
Record Dates: First submitted 2005-12-13; First posted 2005-12-15 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Deep Vein Thrombosis; Pulmonary Embolism; D-dimer; Recurrence; Duration of Anticoagulation; Vitamin K Antagonists
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples for D-dimer assays or other coagulation tests

SUMMARY:
The results of the Prolong study, currently submitted for publication, show that patients with a first unprovoked venous thromboembolic event who have altered D-dimer levels, measured one month after anticoagulation with vitamin K antagonists is stopped, have a high rate of recurrences (about 14%) and a prolongation of anticoagulation is effective in reducing significantly this rate. Those patients with normal D-dimer (about 60% of all patients examined) have a low rate of recurrences (about 5%) and likely a prolongation of anticoagulation in all these patients cannot be recommended.

In line with these results, the Prolong-Two study aims at assessing the predictive role for recurrence of D-dimer levels measured: a) during anticoagulation, b) one month after its withdrawal and c) periodically during follow up.

Patients with a first unprovoked venous thromboembolism (including proximal deep vein thrombosis of a leg and/or pulmonary embolism) which are treated with vitamin K antagonists for not less than 6 months are considered for the study. D-dimer assay is performed during anticoagulation and patients with altered results continue the anticoagulation for 6 more months. Those with normal D-dimer stop the anticoagulant treatment and are again examined one month later. Anticoagulation is resumed for 6 more months in those patients with abnormal D-dimer results but is permanently stopped in those with a normal assay. The latter patients are examined and D-dimer assay performed again every two months to evaluate the natural history of the assay after anticoagulation is stopped and the possible predictive value for recurrence of a change of the assay during follow-up from normal to abnormal results.

ELIGIBILITY:
Inclusion Criteria

* Age > 18 years
* After a first documented idiopathic proximal deep vein thrombosis and/or pulmonary embolism
* After at least 6 months of oral anticoagulation
* After written informed consent

Exclusion Criteria:

* Age > 82 y
* Recurrent venous thromboembolism
* If the Venous thromboembolism occurred:
* during pregnancy or puerperium
* after recent (i.e. within three months) fracture or plaster casting of a leg,
* after immobilization with confinement to bed for three consecutive days after surgery with general anesthesia lasting longer than 30 minutes
* Patients with:
* active cancer
* antiphospholipid antibody syndrome
* antithrombin deficiency
* serious liver disease or renal insufficiency (creatininemia > 2 mg/dL),
* other indications for anticoagulation or contraindications for this treatment
* limited life expectation
* Patients who live too far from the clinical center

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a single previous idiopathic venous thromboembolic event who stop anticoagulation
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2005-08; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gualtiero Palareti, MD, Study Chair — Dept. Angiology & Blood Coagulation, University Hospital S. Orsola-Malpighi, Bologna
Locations (1):
- Dept. Angiology & Blood Coagulation; Azienda Ospedaliero-Universitaria di Bologna, Policlinico S. Orsola-Malpighi, Bologna, BO, Italy

REFERENCES:
- [Derived] Cosmi B, Legnani C, Pengo V, Ghirarduzzi A, Testa S, Poli D, Prisco D, Tripodi A, Palareti G; PROLONG Investigators (on behalf of FCSA, Italian Federation of Anticoagulation Clinics). The influence of factor V Leiden and G20210A prothrombin mutation on the presence of residual vein obstruction after idiopathic deep-vein thrombosis of the lower limbs. Thromb Haemost. 2013 Mar;109(3):510-6. doi: 10.1160/TH12-01-0041. Epub 2013 Jan 10. PMID 23306310
- [Derived] Cosmi B, Legnani C, Tosetto A, Pengo V, Ghirarduzzi A, Testa S, Prisco D, Poli D, Tripodi A, Marongiu F, Palareti G; PROLONG Investigators (on behalf of Italian Federation of Anticoagulation Clinics). Usefulness of repeated D-dimer testing after stopping anticoagulation for a first episode of unprovoked venous thromboembolism: the PROLONG II prospective study. Blood. 2010 Jan 21;115(3):481-8. doi: 10.1182/blood-2009-08-237354. Epub 2009 Nov 16. PMID 19965693
- [Derived] Palareti G, Cosmi B, Legnani C. D-dimer testing to determine the duration of anticoagulant therapy. Curr Opin Pulm Med. 2007 Sep;13(5):393-7. doi: 10.1097/MCP.0b013e3282058b94. PMID 17940483